CLINICAL TRIAL: NCT02628171
Title: Impact of Cashew Nuts in the Human Diet: Measured Energy Value and Effects on Cardiovascular Disease Risk Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Beltsville Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Baer, Research Physiologist, USDA Beltsville Human Nutrition Research Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: HS52
Record Dates: First submitted 2015-10-14; First posted 2015-12-11 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Participants will receive a controlled diet (base diet), typical of an American diet, with 0 g/day of cashew nuts (control).
  Interventions: Other: Base Diet
- Cashew (Active Comparator): Participants will receive a controlled diet, typical of an American diet, with 42 g/day of cashew nuts (base diet with cashew nuts).
  Interventions: Other: Base Diet with Cashew Nuts

INTERVENTIONS:
Other: Base Diet — Participants will receive a controlled diet with 0 g/d of cashew nuts. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Arms: Control
Other: Base Diet with Cashew Nuts — Participants will receive a controlled diet with 42 g/d of cashew nuts. Meals will be prepared using traditional American foods with a macronutrient composition representative of a typical American diet.
  Arms: Cashew

SUMMARY:
This study evaluates the effect of cashew nut consumption on traditional and emerging markers of cardiovascular disease (CVD) risk and determines the usable energy content of a serving of cashew nuts for accurate food labelling.

DETAILED DESCRIPTION:
The cardioprotective effects of nuts have been well documented in the scientific literature; however, most of the research has been done with almonds, walnuts, and pistachios, while studies with cashew nuts are lacking. In addition to the cardiovascular literature, our recent studies measuring the metabolizable energy of nuts have demonstrated that the measured energy value of almonds, pistachios, and walnuts is lower than that predicted using the Atwater factors. However, the measured energy value of cashew nuts is unknown. There are two distinct aims of this study - determining the effects of cashew nut consumption on risk factors of CVD, and determining the energy value of cashew nuts in the human diet. The cardiovascular effects of cashew nuts will be determined by measuring both traditional and emerging risk factors. The metabolizable energy value of cashew nuts will be calculated based on the chemical composition and energy content of the consumed diet and excreta. This will provide a better estimate of the energy value than simply calculating energy value based on Atwater factors.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 20 and 38 kg/m2
* Fasting glucose ≤ 126 mg/dL
* Blood pressure ≤ 160/100 mm Hg

Exclusion Criteria:

* Presence of kidney disease, liver disease, gout, hyperthyroidism, untreated or unstable hypothyroidism, certain cancers, gastrointestinal disease, pancreatic disease, other metabolic diseases, or malabsorption syndromes
* Use of cholesterol lowering medication
* Use of medication to treat hypertension for less than 6 months
* Active cardiovascular disease (such as a heart attack or procedure within the past six months or participation in a cardiac rehabilitation program within the last six months, stroke, or history/treatment for transient ischemic attacks in the past six months, or documented history of pulmonary embolus in the past six months)
* Women who have given birth during the previous 12 months
* Pregnant women or women who plan to become pregnant or become pregnant during the study
* Lactating women
* Type 2 diabetes
* Use of prescription or over-the-counter antiobesity medications or supplements (e.g., phenylpropanolamine, ephedrine, caffeine, during and for at least 6 months prior to the start of the study) or history of a surgical intervention for obesity
* Smokers or other tobacco users (during 6 months prior to the start of the study)
* History of eating disorders or other dietary patterns which are not consistent with the dietary intervention (e.g., vegetarians, very low fat diets, high protein diets)
* Known (self-reported) allergy or adverse reaction to cashew nuts or other nuts
* Unable or unwilling to give informed consent or communicate with study staff
* Self-report of alcohol or substance abuse within the past 12 months and/or current acute treatment or rehabilitation program for these problems (long-term participation in Alcoholics Anonymous is not an exclusion)
* Other medical, psychiatric, or behavioral factors that in the judgment of the Principal Investigator may interfere with study participation or the ability to follow the intervention protocol

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in lipid/lipoprotein profile will be measured in blood | Week 0, end of diet period 1 (week 4), beginning of diet period 2 (week 6), end of diet period 2 (week 10)
  The following will be measured in the blood on 2 consecutive days at the beginning and end of each 4-week diet period: lipids and lipoproteins, apolipoproteins, lipoprotein particle number/size, and proprotein convertase subtilisin/kexin type 9 (PCSK9).
Metabolizable energy will be measured based on energy content of the consumed diet and excreta | Second week of diet period 1 (week 2)
  The measured metabolizable energy value of cashew nuts will be calculated based on the energy content of the consumed diet and excreta.
Metabolizable energy will be measured based on energy content of the consumed diet and excreta | Second week of diet period 2 (week 8)
  The measured metabolizable energy value of cashew nuts will be calculated based on the energy content of the consumed diet and excreta.

SECONDARY OUTCOMES:
Pulse Wave will be measured using Sphygmocor EXCEL | Week 0, end of diet period 1 (week 4), beginning of diet period 2 (week 6), end of diet period 2 (week 10)
  Pulse wave analysis and pulse wave velocity will be conducted.
Markers of vascular health will be measured in blood | Week 0, end of diet period 1 (week 4), beginning of diet period 2 (week 6), end of diet period 2 (week 10)
  Adhesion molecules and endothelin-1 will be measured in the blood.
Digestibility (%) will be calculated as (intake - excreted)/intake | Second week of diet period 1 (week 2), second week of diet period 2 (week 8)
  Fat, protein, and fiber digestibility will be calculated (%) and the effect of cashew nuts on nutrient digestibility (%) will be assessed.
Change in systemic inflammation will be measured in blood | Week 0, end of diet period 1 (week 4), beginning of diet period 2 (week 6), end of diet period 2 (week 10)
  Markers of systemic inflammation will be measured, such as IL-6, TNF-alpha, serum amyloid A, and CRP.
Change in hemostasis will be measured in blood | Week 0, end of diet period 1 (week 4), beginning of diet period 2 (week 6), end of diet period 2 (week 10)
  Fibrinogen and factor VII will be measured in the blood.

CONTACTS AND LOCATIONS:
Locations (1):
- USDA Beltsville Human Nutrition Research Center, Beltsville, Maryland, United States

REFERENCES:
- [Derived] Baer DJ, Novotny JA. Consumption of cashew nuts does not influence blood lipids or other markers of cardiovascular disease in humans: a randomized controlled trial. Am J Clin Nutr. 2019 Feb 1;109(2):269-275. doi: 10.1093/ajcn/nqy242. PMID 30753323